CLINICAL TRIAL: NCT02667288
Title: An Open-Label Study of the Safety of A-101 Solution 40% in Subjects With Seborrheic Keratosis on the Trunk, Extremities and Face.
Brief Title: An Open-Label Safety Study of A-101 Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-101-SEBK-303
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2016-12

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A-101 Solution (Experimental): A-101 Solution 40% administered once
  Interventions: Drug: A-101 Solution

INTERVENTIONS:
Drug: A-101 Solution

SUMMARY:
This is an open-label safety study. During this study, the investigator will identify 4 eligible SK Target Lesions on each subject on the trunk, extremities and face.

DETAILED DESCRIPTION:
This is an open-label safety study. During this study, the investigator will identify 4 eligible SK Target Lesions on each subject on the trunk, extremities and face. The Target Lesions will be treated a maximum of 4 times.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Clinical diagnosis of stable clinically typical seborrheic keratosis
3. Subject has 4 appropriate seborrheic keratosis Target Lesions on the trunk, extremities and face that each are eligible for treatment as defined below:

   * Have a clinically typical appearance
   * Have a PLA of 2 or greater and be a discrete lesion
   * Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   * Not be in an intertriginous fold
   * Not be on the eyelids
   * Not be within 5mm of the orbital rim
   * Not be pedunculated
4. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an active method of birth control for the duration of the study
5. Subject is non-pregnant and non-lactating
6. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of any Target Lesion or which exposes the subject to an unacceptable risk by study participation
7. Subject is willing and able to follow all study instructions and to attend all study visits
8. Subject is able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

1. Subject has clinically atypical and - or rapidly growing seborrheic keratosis lesions
2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Lesser -Trelat)
3. Subject has a current systemic malignancy
4. Subject has used any of the following systemic therapies within the specified period prior to enrollment:

   * Retinoids; 180 days
   * Glucocortico-steroids;
   * Anti-metabolites (e.g., methotrexate);
5. Subject has used any of the following topical therapies within the specified period or in a proximity to any Target Lesion, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   * LASER, light or other energy based therapy (e.g., intense pulsed light, photo-dynamic therapy;
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-flurouracil, or ingenol mebutate;
   * Retinoids;
   * Microdermabrasion or superficial chemical peels;
   * Glucocortico-steroids or antibiotics
6. Subject currently has or has had any of the following within the specified period or in a proximity to any Target Lesion that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   * A cutaneous malignancy;
   * A sunburn; currently
   * A pre-malignancy (e.g., actinic keratosis); currently
   * Body art (e.g., tattoos, piercing, etc.); currently
   * Excessive tan; currently
7. Subject has a history of sensitivity to any of the ingredients in the study medications
8. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
9. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Aclaris Therapeutics, Inc.
Locations (1):
- Aclaris Therapeutics, Inc., Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 Solution: A-101 Solution 40% administered topically for a maximum of 4 treatment visits
  A-101 Solution
Period: Overall Study
Arm/Group | A-101 Solution
Started | 147
Completed | 134
Not Completed | 13
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: ITT Population
Arm/Group | A-101 Solution
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 133
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 138
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Lesion Clearance
Description: Proportion of subjects for whom all target lesions were judged to be clear on the Physician Lesion Assessment (PWA) Scale. The PWA scale is a 4 point scale used by the investigator to assess each subject target SK Lesion.
Time Frame: Study day 148
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Solution
Number analyzed (Participants) | 147
Participants | 16

2. Secondary Outcome: Per Subject Percent of Lesion Clearance
Description: Physician Lesion Assessment (PWA) average Per-Subject Percent of target lesions judged to be clear at Visit 12 in the per protocol population. The PWA scale is a 4 point scale used by the investigator to assess the subject's Target SK lesions.
Time Frame: Day 148
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: percentage of lesions cleared
Arm/Group | A-101 Solution
Number analyzed (Participants) | 142
percentage of lesions cleared | 28.17 (35.34)

ADVERSE EVENTS:
Arm/Group | A-101 Solution
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 14/147
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution (N=147)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Seasonal Allergy (Immune system disorders) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and Investigator agree not to publish the results of this study without the prior written consent of the Sponsor